CLINICAL TRIAL: NCT04043325
Title: Diagnosis of Mycoplasma Pneumoniae Infection With Detection of Specific Antibody-secreting Cells in Community-acquired Pneumonia (CAP) Patients of the Randomised Placebo-controlled Multi-centre Effectiveness Trial of Adjunct Betamethasone Therapy (myKIDS-STEP)
Brief Title: Diagnosis of Mycoplasma Pneumoniae Infection With Detection of Specific Antibody-secreting Cells in Community-acquired Pneumonia (CAP) Patients of the Randomised Placebo-controlled Multi-centre Effectiveness Trial of Adjunct Betamethasone Therapy
Acronym: myKIDS-STEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University Children's Hospital Basel (Other); Ostschweizer Kinderspital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00425
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Enzyme-Linked Immunospot Assay

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal specimen, blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Specific antibody-secreting cell (ASC) enzyme-linked immunspot (ELISpot) assay — Clinical samples (nasopharyngeal swabs and max. 5 ml blood) will be collected from patients enroled in the KIDS-STEP study (NCT03474991; children aged 1-10 years) at enrolment (day 1), at day 3, and at day 28.
  Other Names: Specific enzyme-linked immunosorbent assay (ELISA); Specific polymerase chain reaction (PCR)

SUMMARY:
To compare presence and kinetics of Mycoplasma pneumoniae (Mp)-specific immunoglobulin (Ig) M antibody-secreting cells (ASCs) with Mp DNA and Mp-specific IgM antibodies in patients with community-acquired pneumonia (CAP) of the KIDS-STEP study.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is a common serious infection and a leading cause of hospitalisation in children. Knowledge about the underlying pathogen is a major unmet clinical need, particularly in CAP caused by Mycoplasma pneumoniae (Mp). Timely and reliable identification is critical for initiating effective and tailored antimicrobial treatment. However, determining the causative pathogen of childhood CAP is complicated by the low yield of blood cultures and difficulty obtaining specimens from the lower respiratory tract of children. Therefore, clinicians attempt to detect potential pathogens in upper respiratory tract (URT) specimens, knowing that children carry viruses and bacteria in their URT that may or may not be causative for the current pneumonia episode. Consequently, the interpretation of diagnostic tests performed with URT specimens is limited and may lead to unnecessary antimicrobial prescriptions.

The hurdle in differentiating infection from carriage was documented recently for Mp, a frequently reported pathogen underlying CAP in children worldwide (up to 20-40% during epidemics). Current diagnostic tests, including polymerase chain reaction (PCR) of URT specimens or serology, do not reliable differentiate between Mp infection and carriage. Mp is found in the URT in up to 56% of healthy children. These findings challenge recent epidemiological data indicating Mp as the most common bacterial cause of CAP, in up to 23% of hospitalized U.S. children aged 10-17 years. A ≥4-fold increase in IgG antibody levels is still considered the "gold standard" for diagnosing M. pneumoniae infection, but has low sensitivity when e.g. compared with IgM seroconversion and/or a 2-fold IgM increase. In fact, such a definition is also not helpful in acute clinical management, as it requires acute and convalescent sera.

Circulating antigen-specific B cell responses have been investigated in vaccine studies and demonstrated to be more rapid and shorter lived than antibody responses. After exposure, antigen-specific B cells proliferate and differentiate into antibody-secreting cells (ASCs) and memory B cells. ASCs transiently circulate in the peripheral blood in the first days after an antigen encounter. In a recent observational pilot study of children with CAP and healthy controls, we showed that the detection of Mp-specific immunoglobulin (Ig) M ASCs by enzyme-linked immunospot (ELISpot) assay re-classified 15% of PCR-positive and 12% of IgM-seropositive study participants (https://doi.org/10.1164/rccm.201904-0860LE). Thus, the measurement of specific IgM ASCs by ELISpot assay is an innovative, minimally invasive, and rapid test method that optimises diagnosis of Mp CAP in children.

In view of these promising first results, the aim of this study is to establish the diagnosis of Mp infection by the measurement of Mp-specific ASCs by ELISpot in CAP patients enroled in the randomised placebo-controlled multi-centre effectiveness trial of adjunct betamethasone therapy (KIDS-STEP study, Protocol ID: NCT03474991).

ELIGIBILITY:
Inclusion Criteria:

* At least 12 months of age and younger than 10 years of age
* Body weight between 7 kg and 35 kg
* Admission to hospital (i.e. assignment of an inpatient case number)
* Clinical diagnosis of CAP (according to predefined criteria)
* Parent and/or child (as age-appropriate) willing to accept all possible randomised allocations and to be contacted by telephone weekly up to and including at 4 weeks after randomisation
* Informed consent form for trial participation signed by parent

Exclusion Criteria:

* Presence of local chest complications
* Chronic underlying disease associated with an increased risk of very severe CAP or CAP of unusual aetiology
* Bilateral wheezing without focal chest signs (most likely to represent respiratory tract infection affecting the medium airways, i.e. not pneumonia)
* Inability to tolerate oral medication
* Documented allergy or any other known contraindication to any trial medication
* Subacute or chronic conditions requiring higher betamethasone equivalent or known primary or secondary adrenal insufficiency
* Known diabetes mellitus (type 1)
* Hospitalisation within the last two weeks preceding current admission
* Exposure to systemic corticosteroids with completion of treatment <2 weeks from enrolment (courses of up to 7 days) or <4 weeks from enrolment (courses of >7 days)
* Transfer for any reason to a non-participating hospital directly from the paediatric emergency department
* Parent are unlikely to be able to reliably participate in telephone follow-up because of significant language barriers
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, and other dependent persons.

Ages: 1 Year to 10 Years | Sex: All
Age Groups: Child
Study Population: Children from age 1 year weighing at least 7 kilograms and up to a body weight of 35 kilograms and age below 10 years admitted to the hospital with signs and symptoms of CAP will be considered potentially eligible for participation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Mp-specific IgM ASCs by ELISpot assay | Day 1 (at enrolment)
  Diagnosis of Mp infection in CAP patients of the KIDS-STEP study with the detection of Mp-specific IgM ASCs by ELISpot assay at enrolment (day 1).

SECONDARY OUTCOMES:
No detection of Mp-specific IgM ASCs by ELISpot assay | Day 28
  Longitudinal assessment of levels of Mp-specific IgM ASCs by ELISpot assay.
Detection of Mp-specific DNA by PCR | Day 28
  Longitudinal assessment of levels of Mp-specific DNA by PCR.
Detection of Mp-specific IgM by ELISA | Day 28
  Longitudinal assessment of levels of Mp-specific IgM by ELISA.
Detection of specific IgM ASCs against other pathogens by ELISpot assay | Day 1
  Diagnosis of infection with other respiratory pathogens than Mp in CAP patients of the KIDS-STEP study with the detection of specific IgM ASCs by ELISpot assay at enrolment (day 1).

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No